CLINICAL TRIAL: NCT01332734
Title: Microcirculatory Changes During Open Label Magnesium Sulphate Infusion in Severe Sepsis and Septic Shock
Brief Title: Microcirculatory Changes During Magnesium Sulphate Infusion in Sepsis
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Collaborators: Lithuanian University of Health Sciences (Other)
Responsible Party: Andrius Pranskunas, Lithuanian University of Health Sciences
Other Study IDs: 2010-03.03 nr BE-2-6
Record Dates: First submitted 2011-04-04; First posted 2011-04-11 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: microcirculation; SDF; magnesium sulfate
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Magnesium Sulfate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- severe sepsis and septic shock
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate — 2 gram in 1 hour

SUMMARY:
During infections (sepsis) bloodflow in small vessels (microcirculation) becomes disturbed. Restoration of bloodpressure and cardiac performance may not be sufficient to correct these alterations. Magnesium is a potent vasodilator which may be used to open up the small vessels, in order to reduce organ failure.

DETAILED DESCRIPTION:
In a single-center open label study we evaluated the effects of magnesium sulphate (MgS) infusion on the sublingual microcirculation perfusion in fluid resuscitated patients with severe sepsis and septic shock within the first 48 hours after ICU admission. Directly prior to and after 1 hour of magnesium sulphate (MgS) infusion (2 gram) systemic hemodynamic variables, sublingual SDF images and standard laboratory tests, were obtained.

ELIGIBILITY:
Inclusion Criteria:

* severe sepsis and septic shock

Exclusion Criteria:

* pregnancy
* oral bleeding
* age < 18 years
* liver cirrhosis
* acute arrhythmias
* advanced malignancy or a mean arterial pressure (MAP) < 65 mmHg refractory to vasopressors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: severe sepsis and septic shock after adequate fluid resuscitation according to pulmonary artery catheter measurements
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2010-03; Primary Completion 2010-08 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
microvascular flow index | 1 hour
  Directly prior to and after 1 hour of magnesium sulphate (MgS) infusion (2 gram) systemic hemodynamic variables, sublingual SDF images and standard laboratory tests, were obtained.

CONTACTS AND LOCATIONS:
Overall Officials: A Pranskunas, MD, Principal Investigator — Lithuanian university of sciences
Locations (1):
- Hospital of Lithuanian university of health sciences, Kaunas, Lithuania